CLINICAL TRIAL: NCT05582512
Title: Clinical Characteristics and Long Term Impact on Pediatric COVID-19 in Taiwan
Status: Recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202206053RINC
Record Dates: First submitted 2022-10-10; First posted 2022-10-17 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Long Covid19; COVID-19 Pneumonia; Multisystem Inflammatory Syndrome in Children
Keywords: COVID-19; long COVID; MIS-C
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; pediatric multisystem inflammatory disease, COVID-19 related; COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — Blood, throat or nasopharyngeal swab, stool, sputum, BAL, CSF
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Clinical Characteristics of pediatric COVID-19 by the retrospective research group: Analyze all clinically visible data of hospitalized children with COVID-19 infection (different virus strains), and then find the cause of severe disease and related risk factors for disease
  Interventions: Other: sequelae tracking
- acute case receiving group (including children with multisystem inflammatory syndrome): 1. The correlation between the microbial flora of the respiratory tract and the central nervous system and the severity of SARS-CoV2 pneumonia and host immunity (host inflammatory biomarkers, antibody library/cell receptor library, chemokines, cytokines, cell-regulated immune responses, table Epitope mapping, host transcriptome studies)
  2. To explore the correlation between the clinical manifestations of gastrointestinal tract and liver and SARS-CoV-2 infection and the analysis of gut microbiota
  3. To analyze the host gene factors of COVID-19 patients.
  4. To explore the changes of brain injury biomarkers (Biomarker) in acute and chronic phases, and to analyze the correlation with changes in brain structure and other clinical factors (e.g. severity of neurological symptoms)
  Interventions: Other: sequelae tracking
- children's long COVID-19 tracking group: 1. Clarify the incidence and persistent impact of COVID-19 symptoms in children through outpatient assessment, and further analyze the factors related to preventing the development of COVID-19. / Conduct long-term follow-up through brain MRI and neurophysiological examinations to explore the effects of COVID-19 infection on children brain structure and peripheral nerve function, and analyze the association of risk factors and other clinical symptoms. A psychiatric clinical diagnostic interview was also conducted to establish a psychiatric diagnosis. The emotional and behavioral assessment scale was used to fully evaluate the mental state and family social function.
  2. To analyze the correlation between host genes and antibody repertoire/receptor repertoire, epitope mapping, microbial phase, and prognosis of severe COVID-19 patients
  Interventions: Other: sequelae tracking
- seroepidemiological research group: Through the antibody test and the content of the questionnaire, we can better understand the epidemiology of the COVID-19. Including the proportion of asymptomatic infections, the scale of infection, the speed of transmission, etc. Vaccinated people can also learn about the speed of antibody decline
  Interventions: Other: sequelae tracking
- healthy control group: Provide a sample of the normal population of the "Acute Reception Unit". To carry out respiratory microbial flora, host inflammatory biomarkers, antibody library/receptor library, chemokines, cytokines, cell-mediated immune responses, epitope mapping, brain MRI, neurophysiological examinations (neurophysiological examinations) Conduction, brain waves, sleep watch checks, etc.), brain injury biomarkers (Biomarker), healthy control group studies of host transcriptome
  Interventions: Other: sequelae tracking

INTERVENTIONS:
Other: sequelae tracking — An integrated outpatient clinic for "Long COVID-19 Syndrome in Children" will be established to conduct systematic tracking of body, lung function, nerves and psychology. Children with neurological complications or other confirmed diagnoses will undergo physical, neurological, pulmonary function and brain MRI and neurophysiological examinations, sleep examinations, and conduct psychiatric clinical diagnostic interviews to establish a psychiatric diagnosis. Status and family social function, the intelligence development status was examined by intelligence test, and cognitive function was measured by neuropsychological test. Understand the microbial flora, immune function and incidence of allergic diseases after long-term COVID-19 infection

SUMMARY:
This project will study severe COVID-19 related factors, host genes, biomarkers, and prognosis of severe encephalitis in children, and conduct:

1. Retrospective clinical analysis of children with COVID-19, to analyze the clinical manifestations of children with new crown infection, and to find the relevant factors of severe disease.
2. Prospective acceptance in the acute phase: mainly to understand the correlation between the interaction of host factors, viruses and microorganisms and the severity.
3. Children's long COVID-19 Tracking Team An integrated outpatient clinic for "Long COVID-19 Syndrome in Children" will be established to conduct systematic tracking of body, lung function, nerves and psychology. Children with neurological complications or other confirmed diagnoses will undergo physical, neurological, pulmonary function and brain MRI and neurophysiological examinations, sleep examinations, and conduct psychiatric clinical diagnostic interviews to establish a psychiatric diagnosis. Status and family social function, the intelligence development status was examined by intelligence test, and cognitive function was measured by neuropsychological test. Understand the microbial phase, immune function and incidence of allergic diseases after long-term new coronavirus infection.
4. Seroepidemiological Study Group Exploring the seroepidemiology of different groups of health care workers and non-health care workers will allow us to better understand the magnitude of natural infection among children and age groups in the community and the infection profile of health care workers during this period.

This trial includes multiple groups of prospective cases to explore the impact of the new coronavirus on children and the mechanism of severe illness, and integrates various specialties and branches of the Children's Hospital to conduct a summary trial, which is expected to understand children's new crown and community epidemiology, children infected with new crown Clinical manifestations of the virus, risk factors and effects on various systems, combined with host microbiome, immune function analysis and whole-exome sequencing, to improve the detection of new coronavirus (including long-term new coronary syndrome and pediatric multisystem inflammatory syndrome). Mechanisms of host factors and interactions with microbes to improve outcomes and severe incidence in children.

DETAILED DESCRIPTION:
1. "Clinical Characteristics of pediatric COVID-19）" by the retrospective research group

   * Subject inclusion criteria: COVID-19 positive cases younger than 18 years old from January 1, 2020 to June 13, 2022.
   * Subject exclusion conditions: (none) The number of people to be included is expected to be 3000, and a retrospective case study data collection will be conducted.
2. Prospective case receiving group: divided into four groups: "acute case receiving group" (including children with multisystem inflammatory syndrome), "children's long COVID-19 tracking group", "seroepidemiological research group", "healthy control group" ", in which the "Acute Case Receipt Team" will simultaneously accept cases in Hsinchu and Yunlin Branches.

1. "Acute Receiving Group" (including children with multisystem inflammatory syndrome)

* Subject inclusion conditions: Novel coronavirus positive sick children younger than 18 years old
* Subject exclusion conditions: (none) The above is expected to be included in the number of 200 people will carry out the following (A) Complications caused by new coronavirus infection such as pneumonia (Pneumonia), Multisystem Inflammatory Syndrome in Children (MIS-C), encephalitis (Encephalitis), croup (Croup), sepsis (Sepsis), acute Respiratory distress syndrome (ARDS) and other host gene studies (Host factors) by whole exome sequence (WES).

(B) Testing the respiratory tract, intestinal tract, and central nervous system of 2019-nCoV, microbiota, host inflammatory biomarkers (biomarker: CRP, procalcitonin, DIC profiles…), serum antibody titers and antibody library/ Cell receptor library (spike specific B cell repertoire and T cell repertoire), chemokines (chemokines), cytokines (cytokines: IL-6...), cell-regulated immune response, epitope mapping, immune function test (such as IgG, IgA, IgM, Lymphocyte subset...), host transcriptome research. (see table below) (C) Patients with neurological complications will undergo neurological, pulmonary function, brain MRI and neurophysiological examinations, as well as brain injury biomarkers (Biomarker) changes in acute and chronic phases. (see table below) (D) Physiological monitor of heart rate variability or ECG signal collection over 7 to 14 days and compared with recovery period signal.

(E) Abdominal ultrasound and other tests will be performed for those with abnormal liver function.

(F) Related tests for acute renal failure (CBC+DC, BUN/creatinine/uric acid/Na/K/Cl/LDH/blood gas and urinalysis)

2. "Children's long COVID-19 Tracking Group"

* Subject inclusion conditions: COVID-19 positive cases
* Exclusion conditions for subjects: It is necessary for those who are not suitable to perform "MRI". If there is a metal substance that cannot be removed from the body or a serious disease cannot cooperate with this examination, it is necessary to avoid unexpected occurrences when performing "MRI". Risk considerations, sensory or motor impairments and pregnancy are also inconvenient to perform MRI. For the purpose of the study, those with other causes of encephalitis or those with hypoxic conditions that may affect the cognitive function of the brain are also included in the exclusion conditions in order to avoid errors in the interpretation of the test results.

Exclusions: Anyone who has any of the following conditions cannot participate in this study:

1. You have metal substances that cannot be removed or implanted, such as: braces, metal nails, artificial electronic ears, heartbeat pacemakers, etc. Because of the inability to perform brain MRI, it is not suitable to participate in this trial.
2. Have major physical diseases.
3. Sensory impairment, such as deafness.
4. Movement disorders, such as cerebral palsy.
5. Uncontrolled and stable epilepsy.
6. Pregnant women are not suitable to participate in this test. (If you are pregnant or not sure if you are pregnant, please let the researcher know in advance so that a pregnancy test can be performed).
7. Those who have suffered from hypoxia due to encephalitis or other reasons not caused by enterovirus infection are not suitable to participate in this test.

The number of people expected to be included above is 1,000, and the following will be carried out (A) Establish an integrated outpatient tracking of "Long COVID-19" to conduct systematic tracking of body, lung function, nerves, and psychology. Children with neurological complications or other confirmed diagnoses will undergo physical, neurological, pulmonary function and brain MRI and neurophysiological examinations, sleep examinations, and conduct psychiatric clinical diagnostic interviews to establish a psychiatric diagnosis. Status and family social function, the intelligence development status was examined by intelligence test, and cognitive function was measured by neuropsychological test.

(B) Microbial phase, immune function and incidence of allergic diseases after long-term 2019-nCoV infection.

3. "Seroepidemiological Research Group"

* Subject inclusion conditions:

  1. Voluntarily join the medical staff receiving blood draws. The medical staff of National Taiwan University Hospital, including physicians, nurses, administrative staff, research assistants, cleaning and delivery staff, etc., receive cases in groups according to age. 20-29, 30-39, 40-49, 50-59, and over 60 years old, each group received 60 cases, a total of 300 people. Voluntary participation in non-medical staff receiving blood draws.
  2. The general public who solicited voluntary non-medical workers from the community, received 60 cases in each group of 0-9, 10-19, 20-29, 30-39, 40-49, 50-59, and over 60 years old. people, a total of 420 people.
* Subject exclusion conditions: those who are unwilling to accept blood draws. The above is expected to include 720 people. "Seroepidemiology of novel coronavirus" will be performed, and blood will be drawn three times, once after consent and once after 3 months and 6 months.
* COVID-19 antibody test Serum samples will be tested with commercially available validated test kits, such as Roche's Elecsys Anti-SARS-CoV-2 Assay (Roche Molecular System Inc., CA, USA). Antibodies tested include anti-S and anti-N antibodies. Verify by in-house ELISA or Western blot if necessary.

  4. "Healthy Control Group"
* Inclusion criteria for subjects: "No" healthy individuals with complications after new coronavirus infection or long-term new coronary syndrome Test the respiratory tract and intestinal microbiota (Microbiota), host inflammatory biomarkers, serum antibody titers and antibody library/receptor library of novel coronavirus, chemokines, cytokines, and cell-regulated immunity in healthy control groups Response, epitope mapping, brain MRI, neurophysiological examination (nerve conduction, brain wave, sleep watch examination, etc.), brain injury biomarkers (biomarker), host transcriptome research
* Subject exclusion conditions: (none) The above is expected to include 200 people, and the "acute receiving group" will be matched with the same sex and a normal control group of plus or minus 1 year old.

ELIGIBILITY:
Inclusion Criteria:

* COVID-19 positive cases

Exclusion Criteria:

1. You have metal substances that cannot be removed or implanted, such as: braces, metal nails, artificial electronic ears, heartbeat pacemakers, etc. Because of the inability to perform brain MRI, it is not suitable to participate in this trial.
2. Have major physical diseases.
3. Sensory impairment, such as deafness.
4. Movement disorders, such as cerebral palsy.
5. Uncontrolled and stable epilepsy.
6. Pregnant women are not suitable to participate in this test. (If you are pregnant or not sure if you are pregnant, please let the researcher know in advance so that a pregnancy test can be performed).
7. Those who have suffered from hypoxia due to encephalitis or other reasons not caused by enterovirus infection are not suitable to participate in this test.

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: COVID-19 positive cases younger than 18 years old
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
risk factor and complication | over 3 months
  Clinical symptoms, for example: cough, Headache, rash......etc.
Multidimensional Fatigue Inventory, MFI)-20 | one month
  for long COVID-19 children and family
seropositive rate of COVID-19 | one day
  Anti-SARS-CoV-2 ELISA assay

CONTACTS AND LOCATIONS:
Overall Officials: Luna-Yin Chang, professor, Study Chair — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Chung Cheng District, Taiwan

REFERENCES:
- [Background] Marks KJ, Whitaker M, Agathis NT, Anglin O, Milucky J, Patel K, Pham H, Kirley PD, Kawasaki B, Meek J, Anderson EJ, Weigel A, Kim S, Lynfield R, Ropp SL, Spina NL, Bennett NM, Shiltz E, Sutton M, Talbot HK, Price A, Taylor CA, Havers FP; COVID-NET Surveillance Team. Hospitalization of Infants and Children Aged 0-4 Years with Laboratory-Confirmed COVID-19 - COVID-NET, 14 States, March 2020-February 2022. MMWR Morb Mortal Wkly Rep. 2022 Mar 18;71(11):429-436. doi: 10.15585/mmwr.mm7111e2. PMID 35298458
- [Background] Shi DS, Whitaker M, Marks KJ, Anglin O, Milucky J, Patel K, Pham H, Chai SJ, Kawasaki B, Meek J, Anderson EJ, Weigel A, Henderson J, Lynfield R, Ropp SL, Muse A, Bushey S, Billing LM, Sutton M, Talbot HK, Price A, Taylor CA, Havers FP; COVID-NET Surveillance Team. Hospitalizations of Children Aged 5-11 Years with Laboratory-Confirmed COVID-19 - COVID-NET, 14 States, March 2020-February 2022. MMWR Morb Mortal Wkly Rep. 2022 Apr 22;71(16):574-581. doi: 10.15585/mmwr.mm7116e1. PMID 35446827
- [Background] Sharma S, Agha B, Delgado C, Walson K, Woods C, Gonzalez MD, Jerris R, Sysyn G, Beiter J, Kamidani S, Rostad CA. Croup Associated With SARS-CoV-2: Pediatric Laryngotracheitis During the Omicron Surge. J Pediatric Infect Dis Soc. 2022 Aug 30;11(8):371-374. doi: 10.1093/jpids/piac032. PMID 35512450
- [Background] Brewster RC, Parsons C, Laird-Gion J, Hilker S, Irwin M, Sommerschield A, Michaelis KA, Lam M, Parsons A, Mansbach JM. COVID-19-Associated Croup in Children. Pediatrics. 2022 Jun 1;149(6):e2022056492. doi: 10.1542/peds.2022-056492. No abstract available. PMID 35257175
- [Background] Martin B, DeWitt PE, Russell S, Sanchez-Pinto LN, Haendel MA, Moffitt R, Bennett TD. Acute Upper Airway Disease in Children With the Omicron (B.1.1.529) Variant of SARS-CoV-2-A Report From the US National COVID Cohort Collaborative. JAMA Pediatr. 2022 Aug 1;176(8):819-821. doi: 10.1001/jamapediatrics.2022.1110. PMID 35426941
- [Background] Pongpitakmetha T, Hemachudha P, Rattanawong W, Thanapornsangsuth P, Viswanathan A, Hemachudha T. COVID-19 related acute necrotizing encephalopathy with extremely high interleukin-6 and RANBP2 mutation in a patient with recently immunized inactivated virus vaccine and no pulmonary involvement. BMC Infect Dis. 2022 Jul 23;22(1):640. doi: 10.1186/s12879-022-07610-0. PMID 35870896
- [Background] Asano T, Boisson B, Onodi F, Matuozzo D, Moncada-Velez M, Maglorius Renkilaraj MRL, Zhang P, Meertens L, Bolze A, Materna M, Korniotis S, Gervais A, Talouarn E, Bigio B, Seeleuthner Y, Bilguvar K, Zhang Y, Neehus AL, Ogishi M, Pelham SJ, Le Voyer T, Rosain J, Philippot Q, Soler-Palacin P, Colobran R, Martin-Nalda A, Riviere JG, Tandjaoui-Lambiotte Y, Chaibi K, Shahrooei M, Darazam IA, Olyaei NA, Mansouri D, Hatipoglu N, Palabiyik F, Ozcelik T, Novelli G, Novelli A, Casari G, Aiuti A, Carrera P, Bondesan S, Barzaghi F, Rovere-Querini P, Tresoldi C, Franco JL, Rojas J, Reyes LF, Bustos IG, Arias AA, Morelle G, Christele K, Troya J, Planas-Serra L, Schluter A, Gut M, Pujol A, Allende LM, Rodriguez-Gallego C, Flores C, Cabrera-Marante O, Pleguezuelo DE, de Diego RP, Keles S, Aytekin G, Akcan OM, Bryceson YT, Bergman P, Brodin P, Smole D, Smith CIE, Norlin AC, Campbell TM, Covill LE, Hammarstrom L, Pan-Hammarstrom Q, Abolhassani H, Mane S, Marr N, Ata M, Al Ali F, Khan T, Spaan AN, Dalgard CL, Bonfanti P, Biondi A, Tubiana S, Burdet C, Nussbaum R, Kahn-Kirby A, Snow AL; COVID Human Genetic Effort; COVID-STORM Clinicians; COVID Clinicians; Imagine COVID Group; French COVID Cohort Study Group; CoV-Contact Cohort; Amsterdam UMC Covid-; Biobank; NIAID-USUHS COVID Study Group; Bustamante J, Puel A, Boisson-Dupuis S, Zhang SY, Beziat V, Lifton RP, Bastard P, Notarangelo LD, Abel L, Su HC, Jouanguy E, Amara A, Soumelis V, Cobat A, Zhang Q, Casanova JL. X-linked recessive TLR7 deficiency in ~1% of men under 60 years old with life-threatening COVID-19. Sci Immunol. 2021 Aug 19;6(62):eabl4348. doi: 10.1126/sciimmunol.abl4348. PMID 34413140
- [Background] Chou J, Platt CD, Habiballah S, Nguyen AA, Elkins M, Weeks S, Peters Z, Day-Lewis M, Novak T, Armant M, Williams L, Rockowitz S, Sliz P, Williams DA, Randolph AG, Geha RS; Taking on COVID-19 Together Study Investigators. Mechanisms underlying genetic susceptibility to multisystem inflammatory syndrome in children (MIS-C). J Allergy Clin Immunol. 2021 Sep;148(3):732-738.e1. doi: 10.1016/j.jaci.2021.06.024. Epub 2021 Jul 2. PMID 34224783
- [Background] Kremer S, Lersy F, Anheim M, Merdji H, Schenck M, Oesterle H, Bolognini F, Messie J, Khalil A, Gaudemer A, Carre S, Alleg M, Lecocq C, Schmitt E, Anxionnat R, Zhu F, Jager L, Nesser P, Mba YT, Hmeydia G, Benzakoun J, Oppenheim C, Ferre JC, Maamar A, Carsin-Nicol B, Comby PO, Ricolfi F, Thouant P, Boutet C, Fabre X, Forestier G, de Beaurepaire I, Bornet G, Desal H, Boulouis G, Berge J, Kazemi A, Pyatigorskaya N, Lecler A, Saleme S, Edjlali-Goujon M, Kerleroux B, Constans JM, Zorn PE, Mathieu M, Baloglu S, Ardellier FD, Willaume T, Brisset JC, Caillard S, Collange O, Mertes PM, Schneider F, Fafi-Kremer S, Ohana M, Meziani F, Meyer N, Helms J, Cotton F. Neurologic and neuroimaging findings in patients with COVID-19: A retrospective multicenter study. Neurology. 2020 Sep 29;95(13):e1868-e1882. doi: 10.1212/WNL.0000000000010112. Epub 2020 Jul 17. PMID 32680942
- [Background] LaRovere KL, Riggs BJ, Poussaint TY, Young CC, Newhams MM, Maamari M, Walker TC, Singh AR, Dapul H, Hobbs CV, McLaughlin GE, Son MBF, Maddux AB, Clouser KN, Rowan CM, McGuire JK, Fitzgerald JC, Gertz SJ, Shein SL, Munoz AC, Thomas NJ, Irby K, Levy ER, Staat MA, Tenforde MW, Feldstein LR, Halasa NB, Giuliano JS Jr, Hall MW, Kong M, Carroll CL, Schuster JE, Doymaz S, Loftis LL, Tarquinio KM, Babbitt CJ, Nofziger RA, Kleinman LC, Keenaghan MA, Cvijanovich NZ, Spinella PC, Hume JR, Wellnitz K, Mack EH, Michelson KN, Flori HR, Patel MM, Randolph AG; Overcoming COVID-19 Investigators. Neurologic Involvement in Children and Adolescents Hospitalized in the United States for COVID-19 or Multisystem Inflammatory Syndrome. JAMA Neurol. 2021 May 1;78(5):536-547. doi: 10.1001/jamaneurol.2021.0504. PMID 33666649
- [Background] DeKosky ST, Kochanek PM, Valadka AB, Clark RSB, Chou SH, Au AK, Horvat C, Jha RM, Mannix R, Wisniewski SR, Wintermark M, Rowell SE, Welch RD, Lewis L, House S, Tanzi RE, Smith DR, Vittor AY, Denslow ND, Davis MD, Glushakova OY, Hayes RL. Blood Biomarkers for Detection of Brain Injury in COVID-19 Patients. J Neurotrauma. 2021 Jan 1;38(1):1-43. doi: 10.1089/neu.2020.7332. Epub 2020 Nov 11. PMID 33115334
- [Background] Kanberg N, Ashton NJ, Andersson LM, Yilmaz A, Lindh M, Nilsson S, Price RW, Blennow K, Zetterberg H, Gisslen M. Neurochemical evidence of astrocytic and neuronal injury commonly found in COVID-19. Neurology. 2020 Sep 22;95(12):e1754-e1759. doi: 10.1212/WNL.0000000000010111. Epub 2020 Jun 16. PMID 32546655
- [Background] Buonsenso D, Munblit D, De Rose C, Sinatti D, Ricchiuto A, Carfi A, Valentini P. Preliminary evidence on long COVID in children. Acta Paediatr. 2021 Jul;110(7):2208-2211. doi: 10.1111/apa.15870. Epub 2021 Apr 18. No abstract available. PMID 33835507
- [Background] Kaliyaperumal D, Rk K, Alagesan M, Ramalingam S. Characterization of cardiac autonomic function in COVID-19 using heart rate variability: a hospital based preliminary observational study. J Basic Clin Physiol Pharmacol. 2021 Mar 12;32(3):247-253. doi: 10.1515/jbcpp-2020-0378. PMID 33705614
- [Background] Goldstein B, Fiser DH, Kelly MM, Mickelsen D, Ruttimann U, Pollack MM. Decomplexification in critical illness and injury: relationship between heart rate variability, severity of illness, and outcome. Crit Care Med. 1998 Feb;26(2):352-7. doi: 10.1097/00003246-199802000-00040. PMID 9468175
- [Background] Raina R, Chakraborty R, Mawby I, Agarwal N, Sethi S, Forbes M. Critical analysis of acute kidney injury in pediatric COVID-19 patients in the intensive care unit. Pediatr Nephrol. 2021 Sep;36(9):2627-2638. doi: 10.1007/s00467-021-05084-x. Epub 2021 Apr 29. PMID 33928439
- [Background] Bjornstad EC, Krallman KA, Askenazi D, Zappitelli M, Goldstein SL, Basu RK; SPARC Investigators. Preliminary Assessment of Acute Kidney Injury in Critically Ill Children Associated with SARS-CoV-2 Infection: A Multicenter Cross-Sectional Analysis. Clin J Am Soc Nephrol. 2021 Mar 8;16(3):446-448. doi: 10.2215/CJN.11470720. Epub 2020 Nov 3. No abstract available. PMID 33144276
- [Background] Alabbas A, Kirpalani A, Morgan C, Mammen C, Licht C, Phan V, Wade A, Harvey E, Zappitelli M, Clark EG, Hiremath S, Soroka SD, Wald R, Weir MA, Chanchlani R, Lemaire M. Canadian Association of Paediatric Nephrologists COVID-19 Rapid Response: Guidelines for Management of Acute Kidney Injury in Children. Can J Kidney Health Dis. 2021 Feb 5;8:2054358121990135. doi: 10.1177/2054358121990135. eCollection 2021. PMID 33614056
- [Background] Deep A, Bansal M, Ricci Z. Acute Kidney Injury and Special Considerations during Renal Replacement Therapy in Children with Coronavirus Disease-19: Perspective from the Critical Care Nephrology Section of the European Society of Paediatric and Neonatal Intensive Care. Blood Purif. 2021;50(2):150-160. doi: 10.1159/000509677. Epub 2020 Jul 14. PMID 32663827
- [Background] Kari JA, Shalaby MA, Albanna AS, Alahmadi TS, Alherbish A, Alhasan KA. Acute kidney injury in children with COVID-19: a retrospective study. BMC Nephrol. 2021 May 31;22(1):202. doi: 10.1186/s12882-021-02389-9. PMID 34059010
- [Background] Brodin P, Arditi M. Severe acute hepatitis in children: investigate SARS-CoV-2 superantigens. Lancet Gastroenterol Hepatol. 2022 Jul;7(7):594-595. doi: 10.1016/S2468-1253(22)00166-2. Epub 2022 May 14. No abstract available. PMID 35576952
- [Background] Brodin P. SARS-CoV-2 infections in children: Understanding diverse outcomes. Immunity. 2022 Feb 8;55(2):201-209. doi: 10.1016/j.immuni.2022.01.014. Epub 2022 Jan 20. PMID 35093190
- [Background] Cheng MH, Zhang S, Porritt RA, Noval Rivas M, Paschold L, Willscher E, Binder M, Arditi M, Bahar I. Superantigenic character of an insert unique to SARS-CoV-2 spike supported by skewed TCR repertoire in patients with hyperinflammation. Proc Natl Acad Sci U S A. 2020 Oct 13;117(41):25254-25262. doi: 10.1073/pnas.2010722117. Epub 2020 Sep 28. PMID 32989130
- [Background] Al-Beltagi M, Saeed NK, Bediwy AS, El-Sawaf Y. Paediatric gastrointestinal disorders in SARS-CoV-2 infection: Epidemiological and clinical implications. World J Gastroenterol. 2021 Apr 28;27(16):1716-1727. doi: 10.3748/wjg.v27.i16.1716. PMID 33967552
- [Background] Merzon E, Manor I, Rotem A, Schneider T, Vinker S, Golan Cohen A, Lauden A, Weizman A, Green I. ADHD as a Risk Factor for Infection With Covid-19. J Atten Disord. 2021 Nov;25(13):1783-1790. doi: 10.1177/1087054720943271. Epub 2020 Jul 22. PMID 32697120
- [Background] Colizzi M, Sironi E, Antonini F, Ciceri ML, Bovo C, Zoccante L. Psychosocial and Behavioral Impact of COVID-19 in Autism Spectrum Disorder: An Online Parent Survey. Brain Sci. 2020 Jun 3;10(6):341. doi: 10.3390/brainsci10060341. PMID 32503172
- [Background] Tanaka T, Okamoto S. Increase in suicide following an initial decline during the COVID-19 pandemic in Japan. Nat Hum Behav. 2021 Feb;5(2):229-238. doi: 10.1038/s41562-020-01042-z. Epub 2021 Jan 15. PMID 33452498
- [Background] Moulin F, El-Aarbaoui T, Bustamante JJH, Heron M, Mary-Krause M, Rouquette A, Galera C, Melchior M. Risk and protective factors related to children's symptoms of emotional difficulties and hyperactivity/inattention during the COVID-19-related lockdown in France: results from a community sample. Eur Child Adolesc Psychiatry. 2022 Jul;31(7):1-12. doi: 10.1007/s00787-021-01752-3. Epub 2021 Mar 9. PMID 33751230
- [Background] Zeytinoglu S, Morales S, Lorenzo NE, Chronis-Tuscano A, Degnan KA, Almas AN, Henderson H, Pine DS, Fox NA. A Developmental Pathway From Early Behavioral Inhibition to Young Adults' Anxiety During the COVID-19 Pandemic. J Am Acad Child Adolesc Psychiatry. 2021 Oct;60(10):1300-1308. doi: 10.1016/j.jaac.2021.01.021. Epub 2021 Feb 12. PMID 33582223
- [Background] Wang L, Li D, Pan S, Zhai J, Xia W, Sun C, Zou M. The relationship between 2019-nCoV and psychological distress among parents of children with autism spectrum disorder. Global Health. 2021 Feb 25;17(1):23. doi: 10.1186/s12992-021-00674-8. PMID 33632259